CLINICAL TRIAL: NCT04686864
Title: A Virtual Parent-led Support Group for Parents of Children and Youth With Eating Disorders: A Mixed Methods Feasibility Study Examining Acceptability, Cost and Parent Outcomes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Jennifer Couturier, Dr. Jennifer Couturier, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12703
Record Dates: First submitted 2020-12-15; First posted 2020-12-29 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Eating Disorders
Keywords: eating disorder; parent support group
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Self-Help Groups; Caregivers

STUDY DESIGN:
Intervention Model Description: We studied the implementation of a virtual parent-led peer support group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent Support Group (Experimental): Support and psychoeducation in a group setting for parents who have a child or adolescent with an eating disorder.
  Interventions: Behavioral: Support Group for Caregivers

INTERVENTIONS:
Behavioral: Support Group for Caregivers — Engage parents in the community via this support group, so they can be supported by other parents who "know the system", can advise them on how to proceed, and empower them to help their children. Parents will learn psychoeducation about eating disorders and how to support their children.

SUMMARY:
There is a gap in the literature about the feasibility and implementation of parent-led support groups for parents who have children or adolescents with eating disorders. In this study, we will be observing the experiences of 40 parents in Ontario who will virtually participate in one of 3 parent-led support groups for parents of children and youth with eating disorders. Parents will be expected to attend the virtual sessions twice a month over the course of six months. We hope to evaluate the acceptability, cost, and parental outcomes of the parent-led support groups via surveys before, during, and after the study, as well as using a post-study interview.

ELIGIBILITY:
Inclusion Criteria:

* have the capacity to write, speak and understand English, in order to participate in the sessions
* have access to the internet/computer to participate in the sessions
* must have a child or adolescent with an eating disorder.

Exclusion Criteria:

* don't have the capacity to write, speak and understand English
* don't have access to the internet/computer
* don't have a child or adolescent with an eating disorder

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Change in number of parents who remain in the support group | Baseline and 6 months later
  We will compare the number of parents who initially sign up for the support group to how many parents have stayed in the support group 6 months later.
Number of support groups each parent attends | 6 months after baseline
  We will take note of how many support groups the parent attends in a 6 month period.
Cost | 12 months after baseline
  To assess cost, we will collect data on the costs of the technology, software, and time (of parents and the facilitator).

SECONDARY OUTCOMES:
Change in Carer Burden | Baseline, 3 months, 6 months
  Carer Burden will be assessed using the Eating Disorders Symptom Impact Scale (EDSIS) - a 24 item measure examining the impact of symptoms on parents' lives. Minimum score is 0, maximum score is 96. A higher score indicates that the child's eating disorder symptoms are having a greater impact on their parent (more burdensome).
Change in Carer Needs | Baseline, 3 months, 6 months
  Carer Needs will be assessed using the Carers Needs Assessment Measure (CaNAM), a 47-item questionnaire examining information received about eating disorders, support received from other people and organizations, support for self, and areas where help is needed. The minimum score is 0, the maximum score is 64. A higher score indicates that the carer has received sufficient information and support for themselves and their child.
Change in Parental Self Efficacy and Collaboration | Baseline, 3 months, 6 months
  Parental self-efficacy and collaboration will be assessed using the Patient and Carer Collaboration Scale -C (PACCS), a 33-item questionnaire examining constructs such as hope, self-care and compassion, externalization of the eating disorder, and boundaries. Each question is evaluated on a scale of 0 to 100, where higher values indicate positive collaboration with their child and higher parental self efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Couturier, MD MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicula M, Grennan L, Loewen T, Crews E, Giuliani K, Webb C, Gouveia MR, Couturier J. Virtual parent-led peer support groups for parents of children with eating disorders: A mixed methods feasibility study. Int J Eat Disord. 2023 Nov;56(11):2107-2119. doi: 10.1002/eat.24042. Epub 2023 Aug 14. PMID 37578287
- [Derived] Grennan L, Nicula M, Pellegrini D, Giuliani K, Crews E, Webb C, Gouveia MR, Loewen T, Couturier J. "I'm not alone": a qualitative report of experiences among parents of children with eating disorders attending virtual parent-led peer support groups. J Eat Disord. 2022 Dec 15;10(1):195. doi: 10.1186/s40337-022-00719-2. PMID 36522772